CLINICAL TRIAL: NCT01074359
Title: A Phase 2a, Double Blind, Randomized, Placebo-controlled, 28 Day, Two-arm, Parallel Group Study of A0001 in Patients With the A3243G Mitochondrial DNA Point Mutation and Evidence of Impaired Mitochondrial Function
Brief Title: Safety and Efficacy Study of A0001 in Patients With the A3243G Mitochondrial DNA Point Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for Commercial Reasons. There were no safety issues involved in the decision to terminate the study.
Sponsor: Penwest Pharmaceuticals Co. (Industry)
Responsible Party: Thomas Sciascia, MD/Chief Medical Officer and VP Clinical Operations and Regulatory Affairs, Penwest Pharmaceuticals Co.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEL01
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Neuromuscular Disease
Keywords: A3243G Mitochondrial DNA Point Mutation
MeSH Terms: conditions — Neuromuscular Diseases | interventions — tocopherylquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A0001 (Experimental): A0001 (0.75 g BID)
  Interventions: Drug: A0001 (alpha-tocopherolquinone)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: A0001 (alpha-tocopherolquinone) — 28 days (1.5 g total daily dose) oral A0001 capsules. Treatment taken twice daily with meals.
  Arms: A0001
Drug: Placebo — 28 days of placebo oral capsules. Treatment taken twice daily with meals.
  Arms: Placebo

SUMMARY:
This is a phase 2a, double-blind, placebo-controlled, single-center study. Twenty-one patients who qualify for the study will be randomly assigned to either active drug or placebo. The study will take place at Newcastle University. Patients will have a 66% chance of getting active drug. Patients will be required to take study treatment orally twice a day for 28 days. A baseline visit will occur within 21 days of screening visit. All patients will be followed for 1 week after completion of study or early withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuromuscular symptoms due to the A3243G mitochondrial DNA point mutation
* PCR/ATP ratio of <1.9 following the Cardiac MRS at screening

Exclusion Criteria:

* Any major illness not due to the A3243G mitochondrial DNA point mutation in the past three months or any significant ongoing chronic medical illness, especially significant central nervous neurological disease limiting capacity to carry out the study
* Use of any investigational product within the past 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Improvement in the rate of ATP recovery ("Vmax") in cardiac muscle as measured by 31Phosphorous Magnetic Resonance Spectroscopy (31P-MRS) | Baseline and Day 28

SECONDARY OUTCOMES:
Improvement in cardiac structure and function as measured by Magnetic Resonance Imaging (MRI) | Baseline and Day 28
Exercise tolerance as measured by a 6 minute walk test | Baseline, Day 14 and Day 28
Improvement in the rate of Maximal ATP recovery (Vmax) as measured by 31Phosphorous Magnetic Resonance Spectroscopy (31P-MRS) MRI of calf muscle during a standardized isolated calf muscle procedure of 2 bouts of plantar flexion exercise | Baseline and Day 28
Fasting blood lactate, fasting blood glucose, fasting blood insulin , fasting blood HbA1c levels | Baseline, Day 14 and Day 28
Mitochondrial disease severity (NMDAS) | Baseline and Day 28
Quality of life (SF-36® Health Survey Questionnaire) | Baseline and Day 28
Global impression of clinical severity | Baseline, Day 14 and Day 28
Modified fatigue impact scale | Baseline, Day 14 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Chinnery, Principal Investigator — University of Newcastle Upon-Tyne
Locations (1):
- University of Newcastle upon Tyne, Newcastle, Framlington Place, United Kingdom